CLINICAL TRIAL: NCT01123551
Title: Nebulized Morphine Versus Intravenous Morphine in the Management of Post Traumatic Pain in Emergency Department (ED)
Brief Title: Efficacy Study of Nebulized Morphine and Intravenous Morphine in Post Traumatic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Morphine
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Post Traumatic Pain
Keywords: Nebulized morphine; Intravenous morphine; Post traumatic; Pain; Emergency department
MeSH Terms: conditions — Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulized Morphine (Experimental): After randomization, patients will receive 10 mg of morphine (1ml) diluted in 4 ml normal saline and nebulized with 6 l/mn during 10 min. Nebulization will be repeated systematically 3 times every twenty minutes unless the patient pain was resolved (VAPS 30%). In addition, patients receive a bolus of IV placebo(5 ml normal saline . IV placebo (2 ml) will be repeated every 10 minutes if the objective of analgesia was not reached .
  Interventions: Drug: nebulized morphine; Drug: Intravenous morphine
- Intravenous morphine (Active Comparator): After randomization, patients will receive a bolus of 5 mg of IV morphine (5 ml. Then, 2mg of IV morphine (2ml) will be added every 10 minutes if the objective of analgesia was not reached (VAPS >30%). In addition, normal saline (5ml)is nebulized with 6 l/mn during 10 min and will be repeated systematically every 20 minutes unless the patient's pain was not resolved (VAPS >30%).
  Interventions: Drug: Intravenous morphine

INTERVENTIONS:
Drug: nebulized morphine — After randomization, patients will receive 10 mg of morphine (1ml) diluted in 4 ml normal saline and nebulized with 6 l/mn during 10 min. Nebulization will be repeated systematically 3 times every twenty minutes unless the patient pain was resolved (VAPS 30%). In addition, patients receive a bolus of IV placebo(5 ml normal saline . IV placebo (2 ml) will be repeated every 10 minutes if the objective of analgesia was not reached .
  Arms: Nebulized Morphine
Drug: Intravenous morphine — After randomization, patients will receive a bolus of 5 mg of IV morphine (5 ml. Then, 2mg of IV morphine (2ml) will be added every 10 minutes if the objective of analgesia was not reached (VAPS >30%). In addition, normal saline (5ml)is nebulized with 6 l/mn during 10 min and will be repeated systematically every 20 minutes unless the patient's pain was not resolved (VAPS >30%).

SUMMARY:
In the emergency department, 60% of patients have an acute pain. Appropriate management of acute pain is a public health priority according to who recommendations. Nebulized morphine has been extensively studied in children but less well in adults.

It offers a non-invasive route for systemic drug delivery, more rapid and less invasive than intravenous (IV) method.

ELIGIBILITY:
Inclusion Criteria:

* Post-traumatic pain with visual analog pain scale( VAPS) ≥ 50%
* Age between 8 and 50 years.

Exclusion Criteria:

* Glasgow coma scale (GCS)< 14,
* Severe injury ,
* Hypotension : blood systolic pressure < 90 mmhg,
* Bradypnea < 12 cpm or SaO2< 90%,
* Chronic pain treatment,
* Aspirin or paracetamol treatment within 6 hours of emergency presentation,
* Nasal trauma, rhinitis, nasal obstruction,
* Incapacity to cooperate,
* Opiate allergy,
* Drug addiction,
* Pregnancy, breast feeding,
* Severe renal and liver failure and chronic obstructive pulmonary disease(COPD)

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
1. Resolution rate | one hour
  resolution is defined as VAPS <30%.

SECONDARY OUTCOMES:
rate of side effects | one hour
  Dyspnea, cutaneous rush, vomiting, nausea, pruritus and dizziness.
Resolution time | one hour
  Resolution time is defined as the time between the starting of the protocol and pain decrease to a Visual Analog Scale less than 30%

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Monastir Governorate, Tunisia